CLINICAL TRIAL: NCT05437016
Title: Effectiveness of Functional Rehabilitation With HUBER Platform Compared to a Standard Program, on the Flexion/Extension Ratio of the Spine, in Patients With Non-specific Chronic Low Back Pain
Brief Title: Functional Rehabilitation With HUBER Platform in the Treatment of Non-specific Chronic Low Back Pain.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thibaut Guiraud (Other)
Responsible Party: Sponsor-Investigator, Thibaut Guiraud, Thibaut Guiraud, PhD, Orpea Group
Organization: Orpea Group (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2022-A00885-38
Record Dates: First submitted 2022-06-23; First posted 2022-06-29 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Chronic Low-back Pain
Keywords: isokinetic; physical activity; rehabilitation; HUBER platform
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: monocentric, prospective, randomised, simple blind study (evaluators) with 2 intervention arms (1:1 ratio)
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HUBER rehabilitation group (Experimental): centre-based and will last 6 weeks, with 4 sessions of 2 hours each per week. All the sessions will be supervised by a physiotherapist and will include: 1h of physiotherapy, 30min of balneotherapy and 30min on the HUBER platform to perform exercises
  Interventions: Behavioral: HUBER exercises
- Standard rehabilitation group (Active Comparator): centre-based and will last 6 weeks, with 4 sessions of 2 hours each per week. All the sessions will be supervised by a physiotherapist and will include: 1h of physiotherapy, 30min of balneotherapy and 30min of exercise on cycloergometer.
  Interventions: Behavioral: Standard exercises

INTERVENTIONS:
Behavioral: HUBER exercises — All the exercises involve mobility, flexibility and muscle strengthening exercises. Specifically, these exercises included self-awareness of the lumbo-pelvic-femoral complex and multidirectional mobility of the lumbar spine. We gradually integrated aerobic exercises and muscle strengthening of the lower limbs, trunk and spine extensors with bodyweight exercises. HUBER exercises require the synergistic activation of various muscle groups of the lower limbs, trunk and upper limbs to develop low-high force levels against the handles.
  Arms: HUBER rehabilitation group
Behavioral: Standard exercises — All the exercises involve mobility, flexibility and muscle strengthening exercises. Specifically, these exercises included self-awareness of the lumbo-pelvic-femoral complex and multidirectional mobility of the lumbar spine. We gradually integrated aerobic exercises and muscle strengthening of the lower limbs, trunk and spine extensors with bodyweight exercises.
  Arms: Standard rehabilitation group

SUMMARY:
The objective of this study is to evaluate the effectiveness of centre-based program of 6 weeks with HUBER platform on the spine flexion-to-extension ratio at 60 and 120˚/s, pain and trunk flexibility in individuals with chronic low back pain (CLBP). A total of 70 individuals with Non-specific Chronic Low Back Pain will be randomised into 2 intervention arms (1:1 ratio) that will be blindly evaluated: 1/ standard rehabilitation group and 2/ HUBER rehabilitation group. Both programs are centre-based and will last 6 weeks, with 4 sessions of 2 hours each per week.

DETAILED DESCRIPTION:
The prevalence of chronic low back pain (CLBP) is increasing with age and the prevalence of sedentary lifestyle. According to guidelines, non-pharmacological approaches such as exercise and physical therapy have been proposed in first line treatments along with psychological follow-up and pain medication if needed. The physiotherapy, used in a comprehensive CLBP rehabilitation program, aims to decrease chronic pain and promotes proprioceptive and postural work, as well as spinal mobility, flexibility and muscle strengthening of the spinal area. Isokinetic concentric strength assessment at 60 and 120˚/s is one of the most commonly used criteria to examine the trunk flexors and extensors muscles strength. The objective of this study is therefore to evaluate the effectiveness of an intensive care program with HUBER platform on the spine flexion-to-extension ratio at 60 and 120˚/s measured by Cybex, pain and trunk flexibility in individuals with non-specific CLBP. A total of 70 individuals with CLBP will be randomised into 2 intervention arms (1:1 ratio) that will be blindly evaluated: 1/ standard rehabilitation group and 2/ HUBER rehabilitation group. Both programs are centre-based and will last 6 weeks, with 4 sessions of 2 hours each per week. All the sessions will be supervised by a physiotherapist and will include 1h of physiotherapy, 30min of balneotherapy and 30min of exercise on cycloergometer for the standard rehabilitation group or 30min of exercise on the HUBER platform for the HUBER group. All patients included will benefit from medical monitoring, evaluations and the rehabilitation program set up at the Clinique de Tréboul, Douarnenez, France.

ELIGIBILITY:
Inclusion Criteria:

* people aged between 20 - 55 years old
* with non-specific chronic low back pain (over 3 months)
* with clinical and radiological assessment.

Exclusion Criteria:

* chronic low back pain of specific etiology (trauma, tumor, inflammatory or infectious disease, and radicular syndrome)
* spine with major anatomical deformations
* any contraindication for the rehabilitation program
* surgery less than 3 months and/or receiving treatment with corticosteroids.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-06-23 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in the flexor to extensor ratio measured by Cybex at 60°/s. | Baseline and post-intervention at 6 weeks
  change at 6 weeks from baseline in the flexor to extensor ratio measured by Cybex at 60°/s

SECONDARY OUTCOMES:
Change in the flexor to extensor ratio measured by Cybex at 120°/s. | Baseline and post-intervention at 6 weeks
  change at 6 weeks from baseline in the flexor to extensor ratio measured by Cybex at 60°/s
Change in the peak torque of the extensor muscles of the spine measured by Cybex at 60 and 120°/s. | Baseline and post-intervention at 6 weeks
  change at 6 weeks from baseline in the strength of the extensor muscles of the spine (peak torque at 60°/s and 120°/s concentric)
Change in the peak torque of the flexor muscles of the spine measured by Cybex at 60 and 120°/s. | Baseline and post-intervention at 6 weeks
  change at 6 weeks from baseline in the strength of the flexor muscles of the spine (peak torque at 60°/s and 120°/s concentric)
Change in the hamstring extensibility (Right/Left) (in degrees) | Baseline and post-intervention at 6 weeks
  The patient was lying in the supine position with the contralateral lower limb extended on the table. The therapist then flexed the hip at 90°, brought the knee to extension until their limit (according to the sensations of the patient). An inclinometer was placed on the anterior tibial tuberosity to measure the angle (in degrees) of the popliteal between the tibia and the femur on both legs.
Change in Extensibility of the Psoas (Right/Left) (in degrees) | Baseline and post-intervention at 6 weeks
  the modified Thomas' test was used to measure flexibility of the hip flexors, which included the iliopsoas muscle group. The patient laid on their back, with both legs hanging freely at the edge of the table. First, they achieved a maximum flexion of both knees using both arms to ensure that the lumbar spine is flexed and flat on the table to avoid an anterior tilt of the pelvis. The patient then lowered the tested limb toward the table, whilst the contralateral hip and knee was held in maximal flexion to stabilize the pelvis and flatten out the lumbar lordosis. Once the final position was reached, the inclinometer was placed along the midline of the femur, between the greater trochanter and the lateral femoral condyles (in degrees). The length of the iliopsoas was measured by the angle of the hip flexion.
Change in Extensibility of the Quadriceps (Right/Left) (in cm) | Baseline and post-intervention at 6 weeks
  Ely's test heal-buttock distance was used to measure the flexibility of the quadriceps. The patient laid in prone position. The therapist stood next to the patient, at the side of the leg that is tested. The patient's knee was flexed to bring their heel as close as possible to their buttock. One hand was on the lower back, the other holding the leg at the heel. The closest distance between the heel and the buttock (in cm) was measured. The test is done on both sides for comparison.
Change in the double-lumbar inclinometry in flexion (in degrees) | Baseline and post-intervention at 6 weeks
  Dual inclinometer technique was used to assess spinal. Lumbar range of motion in flexion, extension, right and left lateral flexion.
Change in the double-lumbar inclinometry in extension (in degrees) | Baseline and post-intervention at 6 weeks
  Dual inclinometer technique was used to assess spinal. Lumbar range of motion in flexion, extension, right and left lateral flexion.
Change in the double-lumbar inclinometry in inclination (Right/Left) (in degrees) | Baseline and post-intervention at 6 weeks
  Dual inclinometer technique was used to assess spinal. Lumbar range of motion in flexion, extension, right and left lateral flexion.
Change in the muscular endurance of the trunk and of the lower limbs (in secondes) | Baseline and post-intervention at 6 weeks
  Shirado-Ito test (spinal flexors), Sorensen test (Extensors of the spine), Killy test.
Change in the Score of Pain (Scale from 0 to 10) | Baseline and post-intervention at 6 weeks
  A visual analogue pain scale graded from 0 to 10 was used to quantify the amount of pain that a patient feels from none (0) to an extreme amount of pain (10)
Change in Fear and Avoidance Belief Questionnaire (FABQ) score | Baseline and post-intervention at 6 weeks
  is a self-reported questionnaire which specifically focuses on how a patient's fear avoidance beliefs about physical activity and work may affect and contribute to their low back pain and resulting disability. Sixteen questions scaled from 0 to 6 (higher the score indicates fear avoidance behaviors). The Physical Activity subscale (FABQ-PA) range from 0 to 24 and the Work subscale (FABQ-W) range from 0 to 42.
Change in Oswestry Disability Index questionnaire score | Baseline and post-intervention at 6 weeks
  is a self-completed questionnaire containing ten topics concerning intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel. Each topic category was followed by 6 statements describing different potential scenarios in the patient's life relating to the topic. The patient checked the statement which most closely resembled their situation. Each question was scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability. The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.

CONTACTS AND LOCATIONS:
Overall Officials: Thibaut Guiraud, PhD, Study Director — ORPEA/CLINEA Group
Locations (1):
- CLINEA - Centre de Rééducation fonctionnelle de Treboul, Douarnenez, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] LE Moal V, Tantot M, Mevellec E, Nouy-Trolle I, Lemoine-Josse E, Besnier F, Guiraud T. Rehabilitation therapy using the HUBER platform in chronic non-specific low back pain: a randomized controlled trial. Eur J Phys Rehabil Med. 2023 Oct;59(5):576-585. doi: 10.23736/S1973-9087.23.07998-4. Epub 2023 Sep 22. PMID 37737050